CLINICAL TRIAL: NCT03451539
Title: SHIFTING OF ANESTHESIS PHYSICIANS OUT OF THE INTENSIVE CARE UNIT
Brief Title: OUT OF THE ICU SHIFTING
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7003
Record Dates: First submitted 2018-02-23; First posted 2018-03-01 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Hospital Rapid Response Team Activation
Keywords: Anaesthetist; ICU; Intensif care unit

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Numerous studies dealt with the hospital doctors' work but little is known about the work of ICU doctors, especially concerning the medical time spent outside the Intensive Care Unit (ICU) which is a significant workload that has never been evaluated to date. The main objective of our study was to evaluate the time spent by ICU doctors outside the unit, for the management of their patients during the IHT and for the care of patients in other departments. Secondary objectives were to describe the organization and distribution of medical time outside the intensive care unit.

In this observational study, which took place during 5 years, from January 2012 to December 2016 in the medical ICU of the "Nouvel Hôpital Civil" at the University Hospitals of Strasbourg, every day after the morning medical staff, the anonymized information were collected in a register.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* Physician anesthetist of Intensive Care Unit of new civil hospital in Strasbourg
* Physician anesthetist who has agreed to participate in the study

Exclusion Criteria:

* Refusal to participate in the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All physician anesthetist of Intensive Care Unit of new civil hospital in Strasbourg
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-02-23 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
daily time spent by physicians outside their service | The period from 2012 to 2017 will be examined
  Evaluation of the daily time spent by intensive care physicians outside their department for the care of patients

CONTACTS AND LOCATIONS:
Locations (1):
- Service Reanimation Medicale, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No